CLINICAL TRIAL: NCT00621348
Title: A RCT to Evaluate the Effect of Normal Saline in 5% Dextrose at Maintenance Rate, N/5 Saline in 5% Dextrose at 2/3 Maintenance Rate and N/5 Saline in 5% Dextrose at Maintenance Rate on Incidence of Hyponatremia in Hospitalized Children.
Brief Title: Maintenance Intravenous Fluids in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Dr Rakesh Lodha, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RL-1
Record Dates: First submitted 2008-02-12; First posted 2008-02-22 (Estimated); Results first posted 2011-08-05 (Estimated); Last update posted 2011-08-10 (Estimated); Status verified 2011-08

CONDITIONS: Hyponatremia
Keywords: maintenance fluids; hyponatremia; vasopressin; children
MeSH Terms: conditions — Hyponatremia; Diabetes Insipidus | interventions — Sodium Chloride; Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Isotonic fluid group (Active Comparator): Normal saline in 5% dextrose at standard maintenance rate
  Interventions: Drug: Isotonic fluid
- Fluid restriction group (Active Comparator): Reduced volume (2/3 maintenance rate) of N/5 saline in 5% dextrose
  Interventions: Drug: Hypotonic fluid
- Hypotonic fluid group (Active Comparator): N/5 saline in 5% dextrose at standard maintenance rate
  Interventions: Drug: Hypotonic fluid

INTERVENTIONS:
Drug: Isotonic fluid — 0.9% saline with 5% dextrose at standard maintenance rate
  Other Names: Dextrose normal saline
  Arms: Isotonic fluid group
Drug: Hypotonic fluid — Reduced volume (two thirds of standard maintenance rate) of N/5 saline in 5% dextrose
  Other Names: Hypotonic fluid,; 0.2 % saline in 5 % dextrose
  Arms: Fluid restriction group
Drug: Hypotonic fluid — N/5 saline in 5% dextrose at standard maintenance rate
  Other Names: 0.2 % saline in 5% dextrose
  Arms: Hypotonic fluid group

SUMMARY:
Hyponatraemia arises in between 20% and 45% of sick hospitalized children. An important reason for this high incidence could be use of hypotonic fluids in sick children for maintenance fluid therapy. There are no randomized controlled trials to evaluate the effect of various types of intravenous fluids on the incidence of hyponatremia in sick hospitalized children.

Hypothesis: Use of normal saline in 5% dextrose or reduced (2/3) volume of N/5 saline in 5% dextrose reduces incidence of hyponatremia (serum sodium 130 mmol/L) by two-thirds when compared to N/5 saline in 5% dextrose at standard maintenance rate in hospitalized children receiving intravenous maintenance fluids.

DETAILED DESCRIPTION:
Hyponatraemia arises in between 20% and 45% of sick hospitalized children. An important reason for this high incidence could be use of hypotonic fluids in sick children for maintenance fluid therapy. There are no randomized controlled trials to evaluate the effect of various types of intravenous fluids on the incidence of hyponatremia in sick hospitalized children. We therefore plan to conduct a randomized controlled trial to evaluate the effect of normal saline in 5% dextrose at standard maintenance rate, reduced volume (2/3 maintenance rate) of N/5 saline in 5% dextrose and N/5 saline in 5% dextrose at standard maintenance rate on the incidence of hyponatremia in hospitalized children, aged 3 months- 12 years. To determine serial plasma vasopressin levels in hospitalized children at baseline, 24 hours and 48 hours of intravenous fluid therapy and compare the values in the three fluid regimens.

Study design: Randomized controlled trial. Hospitalized children who fulfill inclusion criteria and not having any of the exclusion criteria will be considered for the enrolment after written informed consent. Venous blood samples will be taken at enrollment for estimation of serum sodium, potassium, chloride, bicarbonate, blood gas, blood sugar, blood urea, serum creatinine, and plasma osmolality. A sample for estimation of plasma vasopressin will be collected at baseline. After randomization into three groups, one group of children will receive N/5 saline in 5% dextrose at standard maintenance rate (100 ml/kg for the first 10 kg of body weight, 50 ml/kg for the next 10 kg, and 20 ml/kg for body weight exceeding 20 kg).The second group of children will receive N/5 saline in 5% dextrose at 2/3 maintenance rate. The third group will receive dextrose normal saline at standard maintenance rate. Serum Na+, K+ and urine Na+, K+ will be estimated every 12 hourly till the patient is on intravenous fluid therapy and 12 hrs after stopping exclusive intravenous maintenance fluids. Serum and urine osmolality will be estimated every 24 hrs by an osmometer. Plasma vasopressin will be estimated in children in the 3 groups at 24, and 48 hours of intravenous fluid therapy.

Children will be weighed every 24 hours. The fluid balance, sodium balance, free water clearance will be calculated in a subset of children.

The study measurements will be carried out only till the time the child is on exclusive intravenous maintenance fluid therapy or 72 hrs of starting the intravenous fluid therapy. The decision to decrease/ stop intravenous fluid therapy will be left to the treating unit.

The primary outcome measure will be incidence of hyponatremia (defined as serum Na+ less than 130 mmol/L).

The secondary outcomes studied will be Plasma vasopressin levels at 24 hr and 48 hours and incidence of hypernatremia.

Sample size: Based on literature review, the incidence of hyponatremia with standard intravenous fluid therapy is approximately 30%. Sample of 72 patients will be needed in each group to demonstrate the decrease in incidence of hyponatremia to 10%, with a beta of 0.2 (Power 80%) and alpha error of 0.05.

Analysis: The data will be analyzed using STATA software. The outcomes (primary and secondary) in the 3 groups will be compared. For continuous variables, t test or Wilcoxon rank-sum test will be used to determine statistical significance. For categorical variables, chi square test will be used.

ELIGIBILITY:
Inclusion Criteria:

* All children (3 months to 12 years) who are admitted to pediatric ward or pediatric ICU, who require exclusive intravenous maintenance fluid therapy for at least 24 hours will be eligible for the study

Exclusion Criteria:

* Children with illness that have primary fluid and electrolyte imbalance such as:

  * Shock: Defined as acute circulatory failure resulting in decreased tissue perfusion and manifesting as altered sensorium, hypothermia (<35oC), tachycardia, prolonged capillary filling time (>3 seconds), hypotension (BP < 5th percentile for age), oliguria (<0.5 ml/kg/hr), hypoxemia, hyperlactatemia, requirement of fluid bolus and/ or vasopressors.
  * Diarrhea and Dehydration: Children presenting with diarrhea and features of dehydration: lethargy, irritability and altered sensorium, thirst, decreased urine output, sunken eyes & dry mucous membranes, loss of skin elasticity.; children with ongoing diarrhea will be excluded even if there is no dehydration.
  * Fluid Overload: Cirrhosis, Congestive heart failure, Acute and Chronic renal failure, Nephrotic syndrome.
* Abnormal serum sodium or Hyperglycemia at Presentation:

  * Hyponatremia : serum sodium < 130 mmol/L.
  * Hypernatremia : serum sodium >150 mmol/L.
  * Hyperglycemia: blood glucose > 180 mg/ dl.
* Severe Protein Energy Malnutrition: Defined as grade III (50-59% of expected weight for age) and grade IV (less than 50% of expected weight for age) as per IAP classification.
* Child who is receiving drugs which cause abnormality in serum sodium such as diuretics, vasopressin, etc.

Ages: 3 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 167 (Actual)
Dates: Start 2006-09; Primary Completion 2008-04 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh Lodha, MD, Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Result] Kannan L, Lodha R, Vivekanandhan S, Bagga A, Kabra SK, Kabra M. Intravenous fluid regimen and hyponatraemia among children: a randomized controlled trial. Pediatr Nephrol. 2010 Nov;25(11):2303-9. doi: 10.1007/s00467-010-1600-4. Epub 2010 Jul 29. PMID 20668885

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment: September 2006 to April 2008 Analysis: May and June 2008 Pediatric ward and Pediatric intensive care unit in a tertiary care referral hospital in North India
Pre-assignment Details: Patients were stratified based on their age in to three groups (age 3 months to 1 year, 1-5 years, 6-12 years) and stratified randomization was used.
Groups:
- Dextrose Normal Saline: Normal saline in 5% dextrose at standard maintenance rate
- Hypotonic Saline: N/5 saline in 5% dextrose at standard maintenance rate
Period: Overall Study
Arm/Group | Dextrose Normal Saline | Fluid Restriction Group | Hypotonic Saline
Started | 58 | 53 | 56
Completed | 58 | 53 | 56
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dextrose Normal Saline | Fluid Restriction Group | Hypotonic Saline | Total
Number analyzed (Participants) | 58 | 53 | 56 | 167
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 58 | 53 | 56 | 167
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 3 (0.44) | 3 (0.36) | 4 (0.28) | 3.33 (0.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 35 | 43 | 114
  Male | 22 | 18 | 13 | 53
Region of Enrollment [Number; unit: participants]
  India | 58 | 53 | 56 | 167

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Hyponatremia (Defined as Serum Sodium Less Than 130 mmol/L)
Time Frame: 72 hrs
Population: 432 patients were eligible. 203 patients were excluded and 62 patients declined consent . Out of 167 patients, 58 patients were randomized to Arm 1, 53 to arm 2 and 56 to arm 3.Intention to treat analysis was used.
Measure: Number; unit: participants
Arm/Group | Dextrose Normal Saline | Fluid Restriction Group | Hypotonic Saline
Number analyzed (Participants) | 58 | 53 | 56
participants | 1 | 2 | 8
Statistical Analysis 1: Comparison: Dextrose Normal Saline vs Fluid Restriction Group vs Hypotonic Saline; The incidence of hospital-acquired hyponatremia with current standard intravenous fluid therapy was approximately 30%. Sample of 72 patients would be needed in each group to demonstrate the decrease in incidence of hyponatremia (defined as plasma sodium< 130 mEq/L) to 10%, with a power of 80 percent and alpha error of 0.05. In view of short study period and feasibility it was planned a priori to enroll at least 50 patients in each treatment limb; Test type: Non-Inferiority or Equivalence — Equivalence analysis; p < 0.05, Fisher Exact — p value was adjusted for multiple comparisons; Risk Ratio (RR) = 0.12, 95% CI 2-sided [0.016 to 0.93], Standard Error of Mean 0 — The risk ratio is for Group A compared with Group C

2. Secondary Outcome: Incidence of Hypernatremia (Serum Sodium >150 mmol/L)
Time Frame: 72 hrs
Population: Intention To Treat analysis
Measure: Number; unit: participants
Arm/Group | Dextrose Normal Saline | Fluid Restriction Group | Hypotonic Saline
Number analyzed (Participants) | 58 | 53 | 56
participants | 2 | 4 | 2

3. Secondary Outcome: Incidence of Symptomatic Hyponatremia
Description: Defined as Hyponatremia (serum sodium < 130 mnol/L)and presence of symptoms attributed to hyponatremia such as altered sensorium, seizure, headache, and vomiting which can not be explained otherwise.
Time Frame: 72 hrs
Measure: Number; unit: participants
Arm/Group | Dextrose Normal Saline | Fluid Restriction Group | Hypotonic Saline
Number analyzed (Participants) | 58 | 53 | 56
participants | 0 | 1 | 0

4. Secondary Outcome: Incidence of Symptomatic Hypernatremia
Description: Symptomatic hypernatremia is defined as serum sodium > 150 mmol/L and the presence of symptoms like altered sensorium, seizure, headache and vomiting not explained otherwise.
Time Frame: 72 hrs
Population: Intention to Treat analysis
Measure: Number; unit: participants
Arm/Group | Dextrose Normal Saline | Fluid Restriction Group | Hypotonic Saline
Number analyzed (Participants) | 58 | 53 | 56
participants | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Dextrose Normal Saline | Fluid Restriction Group | Hypotonic Saline
Serious Adverse Events (participants affected / at risk) | 1/58 | 1/53 | 0/56
Other Adverse Events (participants affected / at risk) | 2/58 | 4/53 | 2/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dextrose Normal Saline (N=58) | Fluid Restriction Group (N=53) | Hypotonic Saline (N=56)
Death or symptomatic hyponatremia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dextrose Normal Saline (N=58) | Fluid Restriction Group (N=53) | Hypotonic Saline (N=56)
Hypernatremia (Renal and urinary disorders) | 2 (2) | 4 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No